CLINICAL TRIAL: NCT04746209
Title: Alpha/Beta T-cell and B-cell Depleted Allogeneic Transplantation (IDE 13641) Followed by Blinatumomab Therapy for High-Risk B-Acute Lymphoblastic Leukemia: A Pilot Study
Brief Title: Blinatumomab After TCR Alpha Beta/CD19 Depleted HCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Amgen (Industry); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Rachel Phelan, Associate Professor, Department of Pediatrics, Division of Hematology/Oncology/BMT, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Blina Part 2
Record Dates: First submitted 2020-09-09; First posted 2021-02-09 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B-cell Childhood Acute Lymphoblastic Leukemia; B-Cell ALL, Childhood
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Alpha/beta T-cell and B-cell Depleted, Myeloablative HCT (Experimental): Patients who are MRD Negative by Flow cytometry but are MRD Positive by High Throughput Sequencing, will receive a myeloablative conditioning regimen which includes total body irradiation (TBI) followed by an alpha/beta T-cell and B-cell depleted transplant. They will also receive a 28 day continuous infusion of blinatumomab starting on Day 100 post-transplant in the absence of significant ongoing GVHD.
  Interventions: Device: Alpha/Beta T-cell and B-cell depleted HCT; Drug: Blinatumomab
- Alpha/beta T-cell and B-cell Depleted, Reduced Intensity HCT (Experimental): Patients who are MRD Negative by Flow cytometry and are MRD Negative by High Throughput Sequencing, will receive a reduced intensity conditioning regimen followed by an alpha/beta T-cell and B-cell depleted transplant. They will also receive a 28 day continuous infusion of blinatumomab starting on Day 100 post-transplant in the absence of significant ongoing GVHD.
  Interventions: Device: Alpha/Beta T-cell and B-cell depleted HCT; Drug: Blinatumomab

INTERVENTIONS:
Device: Alpha/Beta T-cell and B-cell depleted HCT — Device: Alpha/Beta T-cell and B-cell depletion
Drug: Blinatumomab — 28 day continuous infusion given on Day 100 post-HCT if no significant ongoing GVHD
  Other Names: Blincyto

SUMMARY:
This trial will assess the feasibility of alpha/beta T-cell and B-cell depleted allogeneic hematopoietic cell transplantation (HCT) followed by blinatumomab therapy for high-risk B cell acute lymphoblastic leukemia (ALL) as a means of reducing rates of subsequent relapse and improving survival, while also minimizing treatment-related morbidity/ mortality and late effects. The conditioning regimens will be dependent on the patient's minimal residual disease (MRD) status prior to HCT using high throughput sequencing.

DETAILED DESCRIPTION:
This trial evaluates the ability of a biologically active therapy in blinatumomab, an anti-CD19/CD3 bispecific T-cell engager, to further reduce the risk of leukemia relapse following HCT to improve post-HCT outcomes. The investigators will also utilize an alpha-beta T-cell and B-cell depleted graft to reduce the risk of GVHD along with a reduced intensity conditioning regimen without the use of TBI in patients who are minimal residual disease (MRD) negative using high throughput sequencing (HTS) prior to HCT. For those patients who remain HTS-MRD positive, a myeloablative conditioning regimen will be utilized, also followed by blinatumomab. This multi-institutional pilot study will be limited to 25 (estimated 10-15 per stratum) evaluable children, adolescents and young adults with B-ALL, that have experienced a relapse or have high-risk disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-ALL with no evidence of minimal residual disease in the bone marrow by multi-parameter flow cytometry (FC-MRD negative, <0.01%) and meet at least one of the following:

  1. In remission after first relapse or greater (≥ CR2)
  2. Very-high risk biology ALL that is proceeding to HCT in first remission (e.g. Induction failure, Severe-hypodiploidy, Ph-like ALL)
  3. First remission with persistent disease identified as end of consolidation (EOC) MRD > 0.01%.
* Patients must have an available unrelated or haploidentical donor
* Age ≤ 25 years at time of study enrollment
* Karnofsky Performance Status ≥ 60% for patients 16 years and older and Lansky Play Score ≥ 60 for patients under 16 years of age
* Have acceptable organ function as defined within 14 days of study registration: Renal: creatinine clearance or radioisotope GFR ≥ 60 mL/min/1.73m2 Hepatic: ALT < 5 x upper limit of normal (ULN) and total bilirubin ≤ 3 mg/dL Cardiac: left ventricular ejection fraction ≥ 40% by ECHO/MUGA Pulmonary: No evidence of dyspnea at rest. No supplemental oxygen requirement. If measured, carbon monoxide diffusion capacity (DLCO) > 50%. Central Nervous System: Based on clinical exam, no concern for/evidence of active CNS infection. Patients with fully treated prior CNS infections are eligible. Patients with seizure disorders may be enrolled if seizures are well-controlled on anticonvulsant therapy.
* Patients who have experienced their relapse after HCT are eligible, provided they have no evidence of acute or chronic Graft-versus-Host Disease (GVHD) and are off all transplant immune suppression therapy for at least 7-days (e.g. steroids, cyclosporine, tacrolimus). Steroid therapy for non-GVHD and/or non-leukemia therapy is acceptable.
* Immunotherapy: At least 42 days after the completion of any type of immunotherapy aside from blinatumomab (e.g. tumor vaccines or CAR T-cell therapy).
* XRT: Cranial or craniospinal XRT is prohibited during protocol therapy. ≥ 90 days must have elapsed if prior TBI, cranial or craniospinal XRT
* Sexually active females of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment and for 2 months after the completion of blinatumomab therapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment and for 2 months after the completion of blinatumomab therapy.
* Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* All patients enrolled in this study must have been enrolled in the Blinatumomab Bridging Therapy (BBT) Trial

Exclusion Criteria:

* Active extramedullary disease or presence of chloromatous disease.
* Receiving concomitant chemotherapy, radiation therapy; immunotherapy or other anti-cancer therapy for treatment of disease other than is specified in the protocol.
* Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment). Patients with possible fungal infections must have had at least 2 weeks of appropriate anti-fungal antibiotics and be asymptomatic.
* Pregnant or lactating. The agents used in this study are known to be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 7 days prior to registration to rule out pregnancy.
* Known allergy to any chemotherapies or targeted agents included in this protocol.
* Participating in a concomitant Phase 1 or 2 study involving treatment of disease.
* Active malignancy other than B-ALL.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who are able to receive the blinatumomab infusion [Feasibility] | Day +100 post-HCT
  Percentage of patients who are able to receive the blinatumomab infusion at day +100 post-HCT and complete a minimum of 14/28 planned days

SECONDARY OUTCOMES:
Cumulative incidence of treatment-related adverse events [Tolerability] | Day of HCT to Day +180 post-HCT
  As defined by cumulative incidence of treatment-related adverse events of blinatumomab post-HCT
Overall Survival | Day of HCT to 1 year post-HCT
  Defined as the time interval from the date of transplant to death or last follow up
Disease Free Survival | Day of HCT to 1 year post-HCT
  Defined as the time interval from the date of transplant to death or last follow up or disease relapse
Engraftment | Day +100 and +1 year post-HCT
  Defined as the number of patients who achieve ANC > 500/uL for 3 consecutive days
Primary Graft Failure | Day +28 and + 1 year post-HCT
  is defined as failure to achieve ANC > 500/uL by Day +28
Secondary Graft Failure | Day +28 and +1 year post-HCT
  Patients who initially achieve neutrophil engraftment followed by a decline in ANC < 500/uL that is unresponsive to growth factor therapy
Treatment Related Mortality | Day of HCT to Day +100 and 1 year post-HCT
  Defined as death occurring in a patient from causes other than disease relapse or progression
Acute & Chronic GVHD | Day +100, +180 and 1 year post-HCT
  Incidences of Grades 2-4 and Grades 3-4 acute GVHD
Patient Reported Outcomes | Baseline, Day +100, +180, +1 year post-HCT
  PROMIS Pediatric/Parent Proxy Profile 25 (either pediatric self-report if age 8-17 or parent proxy if age 5-8, or both if feasible) or PROMIS-29 Profile if age 18 or older
Length of Stay | Number of days between the day of transplantation, Day 0, and Day +180 post-HCT
  Define by the total number of days a patient spends in the hospital
Persistence of Minimal Residual Disease (MRD) Negativity | Days +28, +100, +180 and +1 year post-HCT
  Number of patients remaining MRD negative by flow cytometry and/or high throughput sequencing
Relapse | Day of HCT to day +180 and 1 year post-HCT
  Cumulative incidence of relapse in all patients

OTHER OUTCOMES:
Analysis of immune cell phenotyping | Days +19, +91, +135 and +180 post-HCT
  Reconstitution of T, B, and NK cell subsets in the peripheral blood will be analyzed by immune cell phenotyping using flow cytometry.
Functional assessment of lymphocyte subsets | Days +19, +91, +135 and +180 post-HCT
  To assess lymphocyte function, peripheral blood mononuclear cells will be co-cultured with stimulator cells in the presence or absence of blinatumomab.
Serum cytokine analysis | Days +19, +91, +135 and +180 post-HCT
  Plasma cytokines will be measured to examine pro and anti-inflammatory cytokines, chemokines and growth factors produced by donor cells during immune reconstitution and GVHD. The plasma cytokines Eotaxin, Eotaxin-3, GM-CSF, IFN-γ, IL-10, IL-12p70, IL-12/IL-23p40, IL-13, IL-15, IL-16, IL-17A, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IP-10, MCP-1, MCP-4, MDC, MIP-1α, MIP-1β, TARC, TNF-α, TNF-β, VEGF-A, and IL-8 will be measured using a multiplex cytokine analyzer where 10 antibodies specific for the above cytokines are attached to a single well providing cytokine capture and immune specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Phelan, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States